CLINICAL TRIAL: NCT02585609
Title: Sleep Quality in Patients With Advanced Cancer. A Comparison of Objective Assessments and Self-reports of Sleep Quality
Brief Title: Sleep Quality in Patients With Advanced Cancer
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Sleep study II
Record Dates: First submitted 2015-10-13; First posted 2015-10-23 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Sleep Disorders; Neoplasms
Keywords: Sleep
MeSH Terms: conditions — Sleep Wake Disorders; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary focus of this clinical study is the objective and subjective measurements of sleep quality in patients with advanced cancer using opioids. It also examines sleep disturbances and associations between sleep quality and symptoms in order to improve symptom management in patients with advanced cancer.

The overall aim of this study is to improve the clinical understanding of sleep quality in patients with advanced cancer using opioids and to improve the understanding of how sleep quality may best be measured in order to improve symptom management.

ELIGIBILITY:
Inclusion Criteria:

* A verified diagnosis of a malignant disease
* Presence of metastatic/disseminated disease
* Regularly scheduled oral, subcutaneous, transdermal or intravenous opioid treatment corresponding to step III at the WHO pain ladder with a duration of treatment not less than 3 days
* Able to comply with all study procedures
* Signed informed consent according to ICH Good Clinical Practice and national/local regulations

Exclusion Criteria:

* Not consenting to participation
* Not mastering the language used at the study centre
* Severe cognitive impairment as judged by the principal investigator
* Any reason why, in the opinion of the investigator, the patient should not participate
* Impaired use of the dominant arm
* Local anatomical illness or abnormalities precluding the use of polysomnography (e.g. facial tumour)
* having received chemotherapy for more than 4 weeks, having received the previous dose less than 5 days ago and receiving the next dose within the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer using opioids (step III on the WHO pain ladder)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
total sleep time | 24 hours
  1 night total sleep measured for comparison by ambulatory polysomnography (PSG), actigraphy and sleep questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Pål Klepstad, md phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Institutt for sirkulasjon og bildediagnostikk, Trondheim, Norway